CLINICAL TRIAL: NCT06811727
Title: CONTinuous Infusion Versus Intermittent Dosing of ceftaZidime/AVIbactam in Critically Ill Patients With Klebsiella Pneumoniae OXA-48 or Pseudomonas Aeruginosa Infections: A Single-centre Randomized Open-label Trial (ZAVICONT)
Brief Title: CONTinuous Infusion Versus Intermittent Dosing of ceftaZidime/AVIbactam in Critically Ill Patients
Acronym: ZAVICONT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ivan Šitum, MD (Other)
Collaborators: UHC Zagreb, Zagreb, Croatia (Other Government); Daniel Lovrić (Unknown); Mirna Momčilović (Unknown)
Responsible Party: Sponsor-Investigator, Ivan Šitum, MD, subinvestigator, Clinical Hospital Centre Zagreb
Organization: Clinical Hospital Centre Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZAVICONT01
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Severe Infection
Keywords: ceftazidime/avibactam; continuous infusion; critically ill; ICU; Klebsiella pneumoniae OXA-48; Pseudomonas aeruginosa
MeSH Terms: conditions — Infections; Critical Illness; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be informed of their group assignment to maintain study integrity. We opted for this study design, which is not fully blinded, for several practical and clinical reasons. First, the dosing regimen of the drug is complex. According to the SmPC, ceftazidime/avibactam is administered as a prolonged infusion over 2 hours every 8 hours. In a placebo-controlled design, all patients would require an additional infusion, either placebo or the active drug, following the initial 2-hour infusion. By not including a placebo, the control group will follow the SmPC dosing regimen (2-hour infusions every 8 hours), while the intervention group will receive the drug as a continuous infusion over 24 hours. Second, the study involves administration in cardiac and cardiac surgery intensive care units, where patients are at a more significant risk of volume overload. The study was designed without a placebo-controlled arm to minimise unnecessary fluid administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuos ceftazidime/avibactam infusion (Experimental): Continuous infusion will include a loading dose of 2 g/0.5 g administered over 2 hours, followed by continuous infusion of 6 g/1.5 g over 24 hours, equivalent to 0.25 g of ceftazidime per hour. The drug reconstitution and dilution process are shown in Figure 2. The final volume of a solution of CZA will be 50 mL, which gives the concentration of ceftazidime 40 mg/mL, with a 4:1 concentration ratio for avibactam (10 mg/mL). The solution will be administered via an infusion syringe with an infusion rate of 6.25 mL/h. Dose adjustments will be applied according to renal function, calculated using the Cockroft-Gault formula
  Interventions: Drug: Continuos ceftazidime/avibactam infusion
- Intermitent dosing as per SMPC (Active Comparator): Intermittent dosing, as outlined in the SmPC, consists of 2 g/0.5 g administered by prolonged infusion over 2 hours every 8 hours. Dose adjustments will be applied according to renal function, calculated using the Cockroft-Gault formula.
  Interventions: Drug: Intermitent dosing as per SMPC

INTERVENTIONS:
Drug: Continuos ceftazidime/avibactam infusion — Continuous infusion will include a loading dose of 2 g/0.5 g administered over 2 hours, followed by continuous infusion of 6 g/1.5 g over 24 hours, equivalent to 0.25 g of ceftazidime per hour. The drug reconstitution and dilution process are shown in Figure 2. The final volume of solution of CZA will be 50 mL, which gives concentration of ceftazidime of 40 mg/mL, with 4:1 concentration ratio for avibactam (10 mg/mL). The solution will be administered via an infusion syringe, with an infusion rate of 6.25 mL/h. Dose adjustments will be applied according to renal function, calculated using Cockroft-Gault formula
  Arms: Continuos ceftazidime/avibactam infusion
Drug: Intermitent dosing as per SMPC — Intermittent dosing, as outlined in the SmPC, consists of 2 g/0.5 g administered by prolonged infusion over 2 hours every 8 hours. Dose adjustments will be applied according to renal function, calculated using Cockroft-Gault formula.
  Arms: Intermitent dosing as per SMPC

SUMMARY:
Ceftazidime/avibactam (CZA) is an essential treatment option for managing infections caused by multidrug-resistant (MDR) gram-negative (G-) bacteria, including Klebsiella pneumoniae OXA-48 and carbapenem-resistant Pseudomonas aeruginosa. Critically ill intensive care unit (ICU) patients frequently exhibit altered pharmacokinetics (PK) of CZA, potentially compromising optimal PK/pharmacodynamic (PD) target attainment with standard dosing regimens. This study compares the efficacy of continuous infusion (CI) versus conventional intermittent dosing (ID) of CZA in critically ill ICU patients with severe infections caused by K. pneumoniae OXA-48 or P. aeruginosa.

This single-centre, randomized, open-label trial will be conducted at a tertiary care hospital within the University Hospital Centre in Zagreb, Croatia, with a 1:1 allocation ratio. One hundred forty critically ill ICU patients requiring CZA treatment will be randomized to receive either ID (2 g/0.5 g every 8 hours over 2 hours) or an equivalent dose in CI (6 g/1.5 g continuously over 24 hours).

The primary outcome is the microbiological success rate. Secondary outcomes include clinical success rate, time to symptom improvement, length of ICU and hospital stay, 28-day all-cause mortality, pathogen recurrence rate, time to weaning from mechanical ventilation, cumulative vasoactive-inotropic score, adverse events, and the ratio of ceftazidime plasma concentration to the pathogen's minimum inhibitory concentration (C/MIC).

This trial seeks to provide evidence on the optimal administration strategy for CZA in critically ill ICU patients with severe infections due to MDR G- pathogens.

ELIGIBILITY:
Inclusion Criteria:

1. General

   1. Age above or equal to 18 years of age.
   2. Able to provide informed consent personally or by his/her next of kin, as requested by the Ethics Committee.
2. Disease-specific

   1. Critically ill patients requiring admission to the intensive care unit (medical or surgical).
   2. Diagnosed with severe infections.
   3. At least one microbiological sample positive for Klebsiella pneumoniae OXA-48 or Pseudomonas aeruginosa.
   4. Requiring a prescription for ceftazidime/avibactam, by clinical judgement

Exclusion Criteria:

1. General

   1. Known or suspected hypersensitivity to ceftazidime/avibactam, excipients, or any other cephalosporin antibacterial agent. Severe hypersensitivity (e.g. anaphylactic reaction, severe skin reaction) to any other β-lactam antibacterial agent (e.g. penicillins, monobactams or carbapenems).
   2. Withdrawal of informed consent.
   3. Age above 85 years of age.
   4. Female who is pregnant or breast-feeding.
   5. Participation (i.e. signed informed consent) in any other interventional clinical trial of an approved or non-approved antibacterial agent within 30 days before screening.
   6. Any disorder which, in the investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.
2. Laboratory values

   1. Severe neutropenia before or during ceftazidime/avibactam administration.
3. Medical conditions

   1. Death within 48 hours following randomization.
   2. Concomitant acquired immunodeficiency syndrome.
   3. Presence or history of malignant neoplasms or in situ carcinomas.
   4. Duration of ceftazidime/avibactam administration is shorter than 72 hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
microbiological success rate | 28 days
  The aim of this study is to investigate efficacy of continuous infusion of ceftazidime/avibactam compared to conventional intermittent dosing, in treating critically ill ICU patients with severe infections caused by Klebsiella pneumoniae OXA-48 or Pseudomonas aeruginosa. The primary outcome of the study is microbiological success rate, defined by proportion of patients in whom the causative pathogen is absent from specimen at the site of infection.

SECONDARY OUTCOMES:
clinical success rate | 28 day
  The clinical success rate is the proportion of patients who achieve clinical cure or clinical improvement evaluated at the end of therapy.
  Clinical cure is the complete resolution of all signs and symptoms, with no evidence of ongoing infection. Clinical improvement is a significant reduction in infection-related signs and symptoms such that the patient demonstrates considerable progress towards recovery.
time to symptoms improvement | 28 day
  Patients who achieve clinical cure or clinical improvement
length of ICU stay | 28 day
  Length of ICU stay is defined as the total number of days from the day of the first CZA administration (study day on 0) until either:
  Discharge from the ICU (if the patient is transferred out of the ICU before day 28) Day 28 (for patients who remain in the ICU beyond this time)
length of hospital stay | 28 day
  Length of hospital stay is defined as the total number of days from the day of the first CZA administration (study day on 0) until either:
  Discharge from the hospital (if the patient is discharged before day 28) Day 28 (for patients who remain hospitalized beyond this time)
all-cause 28-day mortality after ceftazidime/avibactam initiation | 28 day
  All-cause 28-day mortality is defined as death at any point up to and including study day 28. The 28-day mortality rate will be calculated as the number of deaths divided by the total number of patients in the group, expressed as a percentage.
pathogen recurrence rate on day 28 | 28 day
  The pathogen recurrence rate on day 28 is defined as the proportion of patients who have a recurrence of the initial causative pathogen from clinical or surveillance microbiological samples taken by study day 28 after completion of CZA therapy.
time to weaning from mechanical ventilation | 28 days
  time in hours from the start of the trial to the end of mechanical ventilation
cumulative vasoactive-inotropic score (VIS) | 28 day
  The vasoactive-inotropic score is a quantitative measure that evaluates the cumulative effect of vasoactive and inotropic medications. It is calculated using the following formula:
  VIS = dobutamine dose (μg/kg/min) + adrenaline dose (μg/kg/min) x 100 + noradrenaline dose (μg/kg/min) x 100 + vasopressin dose (IU/kg/min) x 10 + angiotensin II dose (ng/kg/min) x 10000 24-hour VIS quantifies the overall cardiovascular support required over 24 hours. The average daily VIS score will be calculated using the following formula: Daily VIS=∑ (VIS for each interval × interval duration (hours)/24 An interval is defined as the period where drug doses remain constant.

OTHER OUTCOMES:
adverse events | 28 day
  Any adverse event that can be attributed to ceftazidime/avibactam
the ratio of ceftazidime plasma concentration to the pathogen's minimum inhibitory concentration (C/MIC) | 28 day
  The ratio of ceftazidime plasma concentration to the pathogen's minimum inhibitory concentration (C/MIC).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Servais H, Tulkens PM. Stability and compatibility of ceftazidime administered by continuous infusion to intensive care patients. Antimicrob Agents Chemother. 2001 Sep;45(9):2643-7. doi: 10.1128/AAC.45.9.2643-2647.2001. PMID 11502544
- [Background] Gatti M, Pea F. Continuous versus intermittent infusion of antibiotics in Gram-negative multidrug-resistant infections. Curr Opin Infect Dis. 2021 Dec 1;34(6):737-747. doi: 10.1097/QCO.0000000000000755. PMID 34261906
- [Background] Adembri C, Novelli A, Nobili S. Some Suggestions from PK/PD Principles to Contain Resistance in the Clinical Setting-Focus on ICU Patients and Gram-Negative Strains. Antibiotics (Basel). 2020 Oct 6;9(10):676. doi: 10.3390/antibiotics9100676. PMID 33036190
- [Background] Lorente L, Jimenez A, Palmero S, Jimenez JJ, Iribarren JL, Santana M, Martin MM, Mora ML. Comparison of clinical cure rates in adults with ventilator-associated pneumonia treated with intravenous ceftazidime administered by continuous or intermittent infusion: a retrospective, nonrandomized, open-label, historical chart review. Clin Ther. 2007 Nov;29(11):2433-9. doi: 10.1016/j.clinthera.2007.11.003. PMID 18158083
- [Background] Gomez CM, Cordingly JJ, Palazzo MG. Altered pharmacokinetics of ceftazidime in critically ill patients. Antimicrob Agents Chemother. 1999 Jul;43(7):1798-802. doi: 10.1128/AAC.43.7.1798. PMID 10390248
- [Background] Muller AE, Punt N, Mouton JW. Optimal exposures of ceftazidime predict the probability of microbiological and clinical outcome in the treatment of nosocomial pneumonia. J Antimicrob Chemother. 2013 Apr;68(4):900-6. doi: 10.1093/jac/dks468. Epub 2012 Nov 28. PMID 23190766
- [Background] Ali A, Imran M, Sial S, Khan A. Effective antibiotic dosing in the presence of resistant strains. PLoS One. 2022 Oct 10;17(10):e0275762. doi: 10.1371/journal.pone.0275762. eCollection 2022. PMID 36215219
- [Background] Ghazi IM, El Nekidy WS. Editorial: Advances in antimicrobial therapy and combating resistance. Front Pharmacol. 2023 Mar 16;14:1170289. doi: 10.3389/fphar.2023.1170289. eCollection 2023. No abstract available. PMID 37007043
- [Background] Batchelder JI, Hare PJ, Mok WWK. Resistance-resistant antibacterial treatment strategies. Front Antibiot. 2023;2:1093156. doi: 10.3389/frabi.2023.1093156. Epub 2023 Jan 30. PMID 36845830
- [Background] Poole K. Pseudomonas aeruginosa: resistance to the max. Front Microbiol. 2011 Apr 5;2:65. doi: 10.3389/fmicb.2011.00065. eCollection 2011. PMID 21747788
- [Background] Bonomo RA, Burd EM, Conly J, Limbago BM, Poirel L, Segre JA, Westblade LF. Carbapenemase-Producing Organisms: A Global Scourge. Clin Infect Dis. 2018 Apr 3;66(8):1290-1297. doi: 10.1093/cid/cix893. PMID 29165604
- [Background] Chen T, Xu H, Chen Y, Ji J, Ying C, Liu Z, Xu H, Zhou K, Xiao Y, Shen P. Identification and Characterization of OXA-232-Producing Sequence Type 231 Multidrug Resistant Klebsiella pneumoniae Strains Causing Bloodstream Infections in China. Microbiol Spectr. 2023 Mar 22;11(2):e0260722. doi: 10.1128/spectrum.02607-22. Online ahead of print. PMID 36946763
- [Background] Garcia-Gonzalez N, Fuster B, Tormo N, Salvador C, Gimeno C, Gonzalez-Candelas F. Genomic analysis of the initial dissemination of carbapenem-resistant Klebsiella pneumoniae clones in a tertiary hospital. Microb Genom. 2023 Jun;9(6):mgen001032. doi: 10.1099/mgen.0.001032. PMID 37272914
- [Background] Ceron S, Salem-Bango Z, Contreras DA, Ranson EL, Yang S. Clinical and Genomic Characterization of Carbapenem-Resistant Klebsiella pneumoniae with Concurrent Production of NDM and OXA-48-like Carbapenemases in Southern California, 2016-2022. Microorganisms. 2023 Jun 30;11(7):1717. doi: 10.3390/microorganisms11071717. PMID 37512889
- [Background] European Medicines Agency (EMA). Summary of Product Characteristics - Zavicefta 2 g/ 0.5 g powder for concentrate for solution for infusion. https://www.ema.europa.eu/en/documents/product-information/zavicefta-epar-product-information_en.pdf. (accessed 9.11.2024.)
- [Derived] Momcilovic M, Situm I, Erceg A, Siroglavic M, Lovric M, Nizic Nodilo L, Hafner A, Lovric J, Turcic P, Fabijanovic D, Marinic A, Nedeljkovic V, Pasalic M, Percin L, Sipus D, Milicic D, Lovric D. Continuous infusion versus intermittent dosing of ceftazidime/avibactam in critically ill patients with Klebsiella pneumoniae OXA-48 or Pseudomonas aeruginosa infections: a single-center randomized open-label trial (ZAVICONT). Rationale and design. Front Pharmacol. 2025 Aug 7;16:1618987. doi: 10.3389/fphar.2025.1618987. eCollection 2025. PMID 40852616